CLINICAL TRIAL: NCT01316406
Title: A Phase II Placebo Controlled, Multicenter Study to Investigate the Safety and Efficacy of ATH008 Cream in Patients With Palmar-Plantar Erythrodysesthesia Syndrome (PPES) Secondary to Capecitabine Therapy.
Brief Title: Safety and Efficacy Placebo Controlled Study of ATH008 Cream in PPES Patients Secondary to Capecitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancell - Advanced In Vitro Cell Technologies, S.A. (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATH008-CLN02
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Palmar-Plantar Erythrodysesthesia Syndrome
Keywords: safety; efficacy; treatment; PPES; Palmar-Plantar Erythrodysesthesia Syndrome; Hand-foot syndrome; capecitabine
MeSH Terms: conditions — Hand-Foot Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ATH008 cream 3% (Experimental): ATH008 cream 3%
  Interventions: Drug: ATH008
- ATH008 cream 8% (Experimental): ATH008 cream 8%
  Interventions: Drug: ATH008
- ATH008 cream placebo (Placebo Comparator): ATH008 cream placebo
  Interventions: Drug: ATH008

INTERVENTIONS:
Drug: ATH008 — The subject will be incorporated in the study and randomised to ATH008 cream 3% or 8% or ATH008 cream placebo
  Other Names: ATH008 cream

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of ATH008 cream in patients with Palmar-Plantar Erythrodysesthesia Syndrome (PPES) secondary to capecitabine therapy. In part I, the safety and plasmatic levels of the active ingredient and its metabolite will allow to determine the most appropriate and beneficial dose for the second part of the study. In Part II, the efficacy of ATH008 cream in reducing the number of patients presenting PPES grade 2/3 secondary to capecitabine therapy following a four times daily application will be tested.

DETAILED DESCRIPTION:
This is a Phase II Placebo Controlled, Multicenter Study that will involve up to 114 patients with Palmar-Plantar Erythrodysesthesia Syndrome (PPES) secondary to capecitabine therapy. Eligible patients will be enrolled into Part I or Part II of the study.

The first part of the study (Part I) is designed

* to demonstrate the safety of ATH008 cream 1%, 3% and 8% and ATH008 cream placebo,
* to determine the plasmatic levels of the active ingredient and its metabolite after repeated doses of ATH008 cream 1%, 3% and 8%, and
* to determine the grade of PPES at Day 1 and Day 21 of ATH008 cream treatment Part I will have four different arms; patients will receive one of the three different doses of drug product (ATH008 cream 1%, ATH008 cream 3% or ATH008 cream 8%) or placebo (ATH008 cream placebo) in repeated doses (twice daily) during a period of 21 days.

Patients will continue to be assessed for safety and pharmacokinetics of active ingredient and its metabolite (Pre-dose, Day 1 and Day 21). Results of Part I will determine the most appropriate and beneficial dose for the second part of the study.

The second part of the study (Part II) is aimed at demonstrating the safety and efficacy of ATH008 cream in reducing the number of patients presenting PPES grade 2/3 secondary to capecitabine therapy following a four times daily application.

Part II will have three different arms; patients will receive ATH008 cream 3%, 8% or placebo in repeated doses (four times per day) since appearance of PPES grade 1 until appearance of grade 2-3 or a maximum of 4 cycles. Patients will continue to be assessed for safety. The clinical signs will be reported by iconographic register of lesions and pain will be evaluated using a pain scale. Patient will fill a questionnaire reporting QoL.

ELIGIBILITY:
Inclusion Criteria:

* Are under capecitabine monotherapy for treatment of colon or breast cancer at a regimen of 2 weeks on and 1 week off (14+7) and a daily doses between 2000 and 2500 mg/m2.
* Diagnosis of PPES grade 1 in any hand or foot according to the NCI CTCAE v4.03 definition.
* In Part I, subjects still have to undergo at least 1 planned cycle with capecitabine monotherapy.
* In Part II, subjects still have to undergo at least 2 planned cycles with capecitabine monotherapy.

Exclusion Criteria:

* Are younger than 18 years.
* Use of other chemotherapies for the treatment of cancer except trastuzumab (Herceptin®) or bevacizumab (Avastin®).
* Diagnosis of PPES grade 1 in any hand or foot according to the NCI CTCAE v4.03 definition for more than 2 cycles previously to inclusion in this clinical study.
* Have neurologic symptoms greater than grade 1, which under the criteria of the clinician could interfere with PPES diagnosis or study treatment (e.g. hands or feet neuropathy).
* Have any dermatologic condition that in the opinion of the investigator may affect hands or feet or may complicate evaluation during study treatment (e.g. neurodermatitis, psoriasis, etc).
* Have onycholysis with a non-stable grade 1 or onycholysis greater than grade 1 (nail loss, NCI CTCAE v4.03 criteria) which in the assessment of the clinician could interfere with PPES diagnosis or study treatment.
* Need to use other emollient creams or other topical treatments in hands and/or feet during the study.
* Are receiving radiotherapy.
* Have received topical corticosteroids in hands or feet 7 days prior to planned inclusion in the study.
* Are participating in any other investigational studies for the treatment of PPES.
* Have participated in any other investigational studies for the treatment of PPES, or received an experimental therapeutic procedure, considered to potentially interfere with the study in the 4 weeks preceding Day 1.

The above is not a complete list of eligibility criteria. Please see your study doctor for more information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of ATH008 cream in reducing the number of subjects presenting PPES grade 2/3 secondary to capecitabine therapy | minimum every 21 days, maximum of 4 capecitabine cycles, followed by a safety observation period of 14 days
  percentage of subjects that develop PPES grade 2 or 3 according to the NCI CTCAE v4.03 criteria
Safety of ATH008 cream in patients presenting PPES secondary to capecitabine therapy | minimum every 21 days, maximum of 4 capecitabine cycles, followed by a safety observation period of 14 days
  adverse events and serious adverse events (incidence, causality, and severity) related to treatment with ATH008 cream
Plasmatic levels of ATH008 cream when given topically | blood sampling at specific timepoints (Pre-dose, Day 1 and Day 21)
  plasmatic levels of the active ingredient and its metabolite when given topically

SECONDARY OUTCOMES:
Efficacy of ATH008 cream in improving the quality of life of patients presenting PPES | minimum every 21 days, maximum of 4 capecitabine cycles, followed by a safety observation period of 14 days
  quality of life compared to baseline
Efficacy of ATH008 cream in improving signs and symptoms of PPES | minimum every 21 days, maximum of 4 capecitabine cycles, followed by a safety observation period of 14 days
  proportion of subjects that present no PPES signs or symptoms, time to progression and time to improvement of PPES grades,assessment from photographs of erythema, desquamation, existence of blisters, fissures and ulcers; percentage of palms and soles affected by PPES
Assessment of patient reported pain | minimum every 21 days, maximum of 4 capecitabine cycles, followed by a safety observation period of 14 days
  assessment of pain, using a 0-10 score, analysed comparing the values measured during the study treatment period with the baseline pain value
Accumulated dose intensity of capecitabine before and during ATH008 cream treatment | minimum every 21 days, maximum of 4 capecitabine cycles, followed by a safety observation period of 14 days
  accumulated capecitabine dose during study treatment (mg / m2) from the starting of ATH008 cream treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. A. Awada, Principal Investigator — Jules Bordet Institute
Locations (26):
- Belgium (3):
  - Imelda, Bonheiden
  - Institute Jules Bordet, Brussels
  - AZ Maria Middelares, St-Niklaas
- Germany (4):
  - Iniversitätsklinikum Hamburg Eppendorf, Hamburg
  - OncoResearch Lerchenfeld UG, Hamburg
  - Klinikum Offenbach GmbH, Offenbach
  - Prosper Hospital, Recklinghausen
- Italy (4):
  - IRCCS - Istituto Europeo di Oncologia (IEO) di Milano, Milan, Dr. Franco Nolè
  - A.O. Universitaria Policlinico S.Orsola-Malpighi di Bologna, Bologna
  - Azienda Ospedaliero Universitaria "Maggiore Della Carità" di Novara, Novara
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
- Spain (15):
  - Institut Català d'Oncología, L'Hospitalet de Llobregat, Barcelona
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - HGU Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Complejo Hospitalario Regional Reina Sofia, Córdoba
  - Hospital General de Elche, Elche
  - Hospital Clínic i Provincial, Madrid
  - Hospital Gregorio Marañón, Madrid
  - HGU La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital de Navarra, Pamplona
  - Hospital de Torrevieja, Torrevieja
  - Institut Valencià d'Oncologia, Valencia
  - Hospital Miguel Servet, Zaragoza